CLINICAL TRIAL: NCT03656731
Title: Exercise in Older Women With Breast Cancer During Systemic Therapy - a Randomized Controlled Trial (Breast Cancer Exercise Study)
Brief Title: Exercise in Older Women With Breast Cancer During Systemic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Cecilia Margareta Lund, MD, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BREACE
Record Dates: First submitted 2018-08-22; First posted 2018-09-04 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: exercise; older; resistance training; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to the intervention group and control group
Who Masked: Outcomes Assessor
Masking Description: All physical tests will be conducted by masked health care professionals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (n=50) (Experimental): Patients in the intervention group will receive standard care and a 12-week exercise-based intervention.
  Interventions: Other: Breast cancer exercise intervention
- Control group (n=50) (No Intervention): Patient in the control group will receive standard care.

INTERVENTIONS:
Other: Breast cancer exercise intervention — The exercise-based intervention is comprised of:
  1. Supervised and group-based exercise training at the hospital setting two times a week. Each session will last approximately 60 minutes.The program consists of warm-up, exercises for balance and flexibility, progressive resistance training (seven resistance training exercises targeting the large muscle groups), and stretching and relaxation.
  2. Home-based walking with activity tracker assessment. Evaluation and goal-setting in relation to activity (step counts) will be conducted once weekly.
  3. Serving of a protein supplement (protein drink or bar) after each supervised training session.
  Arms: Intervention group (n=50)

SUMMARY:
BREACE is a prospective randomized controlled trial. The aim is to investigate the effect of an exercise-based intervention among older participants with breast cancer treated with adjuvant or first-line systemic therapy.

The hypotheses: That the intervention will maintain or increase physical function levels, reduce symptoms and side effects, improve quality of life and psychological wellbeing, and prevent weight loss and muscle wasting

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* Be operated for primary breast cancer within 12 weeks or
* Be diagnosed with locally advanced or metastatic breast cancer. Be treated with (neo)adjuvant or first or second-line palliative therapy defined as chemotherapy ± HER2 directed treatment, ± antihormonal treatment, antihormonal treatment ± HER 2, directed treatment ± CDK 4/6 inhibitor.
* Be ≥ 65 years of age at the time of signing the informed consent form
* Have an Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2
* Be able to speak and read Danish, and to provide a signed informed consent form.

Exclusion Criteria:

Participants with:

* Any physical condition that hinder the execution of physical exercise training
* Other types of cancer
* Documented and uncontrolled brain metastases that hinder participation in an exercise-based trial, based on the referring oncologist's assessment
* Dementia, psychotic disorders, or other cognitive diseases or conditions that hinder written consent
* Unstable medical disease or history of serious or concurrent illness; any medical condition that might be aggravated by exercise training or that cannot be controlled, including, but not restricted congestive heart failure (NYHA class III-IV), unstable angina pectoris, implantable cardioverter defibrillator (ICD), or myocardial infarction within 6 months, based on the referring oncologist's assessment.

In patients with documented bone metastases:

- A bone metastatic burden or location that poses a risk of injury in the performance of exercise training, as assessed by the referring oncologist.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in the 30-second chair stand test | baseline, 6 weeks, 12 weeks and 24 weeks
  To measure change over time in the lower extremity strength, the number of stands a participant can complete in 30-seconds from a seated position with their arms crossed over the chest, is registered.

SECONDARY OUTCOMES:
The 6-meter Gait Speed Test | baseline, 6 weeks, 12 weeks and 24 weeks
  To asses physical performance at normal and maximal gait speed. The assessment will be conducted by blinded physiotherapist.
The 10-meter Gait Speed Test | baseline, 6 weeks, 12 weeks and 24 weeks
  To asses physical performance at normal and maximal gait speed. The assessment will be conducted by blinded physiotherapist
The 6-minute-walk-test | baseline, 6 weeks, 12 weeks and 24 weeks
  To measure physical capacity and endurance. The distance (measured in meters) a participant is able to walk over a total of six minutes on a hard flat surface. The assessments will be conducted by a blinded physiotherapist
The Handgrip Strength Test | baseline, 6 weeks, 12 weeks and 24 weeks
  Physical function of the upper body will be measured using hand-held dynamometer. The assessment will be conducted by blinded physiotherapist
Stair climb test | baseline, 6 weeks, 12 weeks and 24 weeks
  To measure lower extremity muscle power. The patient will climb a flight of stairs (20 steps) as fast as possible. The assessment will be conducted by blinded physiotherapist.
Adherence to exercise sessions | Up to 12 weeks
  Number of exercise sessions attended out of planned sessions
Physical activity level | baseline and 12 weeks
  Data of step counts will be assessed daily for participants in the intervention group and will be measured with an activity tracker.
European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 | baseline, 6 weeks, 12 weeks and 24 weeks
  Measure quality of life with the EORTC QLQ-C30 patient questionnaire. The questionnaire comprises 30 items, is designed to be cancer specific, and consists of six functional scales (physical, role, cognitive, emotional, social functioning, and global QOL) and symptom scales (fatigue, nausea/vomiting, sleep disturbance, constipation, diarrhea, appetite loss, dyspnea).
European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire BR23 | baseline, 6 weeks, 12 weeks and 24 weeks
  Measure quality of life with the EORTC QLQ-BR23 patient questionnaire. The questionnaire is a breast cancer specific module to EORTC-QLQ-C30, comprises 23 items and consist of functional scales and symptom scales. Each item is scored on a scale from 1 to 4. 1 being "not at all" and 4 being "very much".
M.D. Anderson Symptom Inventory (MDASI) | baseline, 6 weeks, 12 weeks and 24 weeks
  The MDASI patient questionnaire measures the severity of symptoms and the interference with daily living asses by the participant based on the last 24 hours. The questionnaire consist of 13 core symptom items representing symptoms that have been found to have the highest frequency and/or severity among cancer patients with various cancers and treatment types, and 6 interference items representing commonly experienced symptom interference with daily activities.
Hospital Anxiety and Depression Scale (HADS) | baseline, 6 weeks, 12 weeks and 16 weeks
  Measure symptoms of depression and anxiety with the HADS patient questionnaire. The questionnaire comprises a total of 14 items, generates ordinal data, and is designed to measure general anxiety and depression by self-administration. Seven of the items relate to anxiety and seven relate to depression. Each item is scored on a scale from 0 to 3 and this mean a participant can score between 0 and 21 for either anxiety and depression. Scores categorized as follows: normal 0-7, mild 8-10, moderate 11-14, and severe 15-21.
Common Toxicity Criteria for Adverse Events version 4 | up to 6 months
  Number of participants with side-effects to oncological treatment assessed with the Common Toxicity Criteria for Adverse Events version 4. Data will be collected from medical records.
Body weight | baseline, 6 weeks, 12 weeks and 24 weeks
  Weight will be assessed using standard procedures (no shoes, light clothing) and will be reported in kilograms
Body mass index | baseline, 6 weeks, 12 weeks and 24 weeks
  Reported in kg/m^2
whole-body lean body mass (LBM) | baseline and 12 weeks
  Measured with bioimpedance and DXA scans
whole-body fat mass | baseline and 12 weeks
  Measured with bioimpedance and DXA scans
whole-body mineral density | baseline and 12 weeks
  Measured with bioimpedance and DXA scans
Inflammation | Data will be recorded from the medical records
  Inflammatory biomarkers: c-reactive protein, interleukin 6, YKL-40, GDF11 and GDF15.
Number of hospitals admissions | up to 6 months
  Data will be collected from medical records
Causes of hospitalizations | up to 6 months
  Data will be collected from medical records
Lengths of hospitalizations | up to 6 months
  Data will be collected from medical records
Survival | up to 6 months
  Incidences of deaths (cancer-related and other cause) will be registered. The purpose is to investigate whether the intervention may affect survival time/mortality. Data will be collected from medical records.
Adverse events | up to 12 weeks
  Cases of exercise-related injuries or events, including, but not restricted to musculoskeletal-related events, falls, fall-related injuries, bleedings, or cardiovascular events.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev and Gentofte Hospital, Herlev, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen HH, Mikkelsen MK, Lundager I, Lund CM, Johansen JS, Vinther A, Bogh Juhl C, Zerahn B, Ragle AM, Nielsen DL. Exercise in older women with breast cancer during systemic therapy: study protocol of a randomised controlled trial (BREACE). BMJ Open. 2020 Oct 7;10(10):e038674. doi: 10.1136/bmjopen-2020-038674. PMID 33033025

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT03656731/Prot_SAP_000.pdf